CLINICAL TRIAL: NCT05615805
Title: The Effect of Ocular Rinse Volume on Surface Irritation After Povidone-iodine Preparation for Intravitreal Injections: A Randomized Controlled Trial
Brief Title: The Effect of Ocular Rinse Volume on Surface Irritation After Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB #9810
Record Dates: First submitted 2022-10-26; First posted 2022-11-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Intravitreal Injection; Ocular Rinse; Age-Related Macular Degeneration; Diabetic Macular Edema; Cystoid Macular Edema
MeSH Terms: conditions — Macular Degeneration; Macular Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3-mL washout with saline based ocular rinse post injection (Experimental)
  Interventions: Other: OSDI questionnaire; Other: SPEEDII questionnaire
- 10-mL washout with saline based ocular rinse post injection (Experimental)
  Interventions: Other: OSDI questionnaire; Other: SPEEDII questionnaire
- 15-mL washout with saline based ocular rinse post injection (Experimental)
  Interventions: Other: OSDI questionnaire; Other: SPEEDII questionnaire

INTERVENTIONS:
Other: OSDI questionnaire — Ocular Surface Disease Index
Other: SPEEDII questionnaire — Standardized Patient Evaluation of Eye Dryness II questionnaire

SUMMARY:
This is the first randomized controlled trial looking into post-injection rinse volume of standard ophthalmic eyewash and its affect on patient comfort up to 72 hours after injections.

DETAILED DESCRIPTION:
Purpose To evaluate whether the volume of wash out rinse after povidone iodine (PI) application for intravitreal injections (IVI) affects patients' ocular surface irritation.

Methods This was a prospective, single-masked, randomized-controlled trial consisting of 142 subjects . A total of 51, 45, and 46 patients received 3-mL, 10-mL, and 15-mL of ocular rinse respectively. Reductions in the Ocular Surface Disease Index (OSDI) and the Standardized Patient Evaluation of Eye Dryness II (SPEED II) surveys, conducted before and at 24-72 hours post-injection, were analyzed.

ELIGIBILITY:
Inclusion Criteria:

choroidal neovascular membrane or cystoid macular edema requiring intravitreal injections for treatment.

Exclusion Criteria:

active ocular infection, eyelid trauma, graft versus host disease, thyroid eye disease, pregnancy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | 24-72 hours after injection
  Patient symptoms questionnaire, range 0-28, higher score is associated with worse outcome.

SECONDARY OUTCOMES:
Standardized Patient Evaluation of Eye Dryness II | 24-72 hours after injection
  Patient symptoms questionnaire, range 0-48, higher score is associated with worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Dean McGee Eye Institute, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided
Depending on their required use of the data